CLINICAL TRIAL: NCT03176303
Title: A Multi-Center, Open-Label, Prospective Study of SpinalStim™ (MOP-SS) as Adjunctive Care Following Lumbar Fusion Surgery
Brief Title: Study Using the SpinalStim Device Following Lumbar Fusion Surgery
Status: Completed | Type: Observational
Sponsor: Orthofix Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-1702SSPM
Record Dates: First submitted 2017-04-27; First posted 2017-06-05 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Lumbar Spine Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

GROUPS / COHORTS (1):
- Pulsed Electromagnetic Field: one group all of whom will be treated with the PEMF device
  Interventions: Device: SpinalStim

INTERVENTIONS:
Device: SpinalStim — PEMF osteogenesis stimulator

SUMMARY:
This study examines the effect of adjunctive use of the SpinalStim bone growth stimulator on lumbar fusion rate in high risk subjects who have had lumbar fusion surgery. All participants will wear the bone growth stimulator for a minimum of 2 hours/day for 6 months.

DETAILED DESCRIPTION:
The purpose of this post market prospective study is to examine the effect of the adjunctive use of the Orthofix SpinalStim™ device on lumbar fusion rate in high risk subjects who have undergone lumbar fusion surgery. High risk subjects are those who are currently using nicotine, who are having a multi-level fusion, who have had a prior failed fusion at any lumbar level, who are diabetic or who are osteoporotic. Because this is a post market prospective study, subjects who are enrolled in this study will be identified by the Investigator as needing lumbar fusion surgery and asked if they would like to participate in a study looking at the efficacy of lumbar fusion with adjunctive use of the SpinalStim bone growth simulator. The type of lumbar fusion surgery performed (lateral lumbar interbody fusion [XLIF], posterior lumbar interbody fusion [PLIF], anterior lumbar interbody fusion [ALIF], posterolateral fusion) is up to the Investigator; the subjects in the study must be agreeable to using the bone growth stimulator daily for 6 months post surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥ 18 years of age at the time of Informed Consent
2. Requires a lumbar fusion surgery within 30 days of signing Informed Consent.

   a. Surgical approach is according to physician's discretion.
3. Subject has one or more risk factors:

   * Is currently using nicotine
   * multi-level lumbar fusion surgery planned
   * Prior failed fusion at any lumbar level
   * Subject reported diabetes
   * Subject reported osteoporosis
4. Body mass index ≤ 45 kg/m2 at the time of consent.
5. Must have reliable access to an iPhone or an iPad with Wi-Fi access for downloading the free device-specific app (iPhone 5S or higher, iPad, iPad Pro, iPad mini or iTouch using iOS v9.3 or later). When the android version of the mobile app for the SpinalStim becomes available (estimated to be Dec. 2017), subjects who have reliable access to devices using android operating systems will be eligible for study inclusion.
6. Able and willing to complete electronic questionnaires and able to read and understand study instructions in English
7. Able and willing to comply with the study plan and able to understand and sign the study-specific ICF.

Exclusion Criteria:

1. Scoliosis greater than 30 degrees
2. Current alcoholism or drug abuse, and/or any known current addiction to pain medications or medical marijuana
3. Any active malignancy or prior history of malignancy within last 5 years prior to fusion (except basal cell carcinoma of the skin).
4. Any clinically significant finding that places the subject at health risk, impacts the study, or affects completion of the study, in the opinion of the Investigator
5. Any psychiatric illness that prevents subject from completing the assessments accurately, in the opinion of the Investigator
6. Prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects from all over the United States are eligible for enrollment as long as they meet the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
fusion rate | 12 months
  number of subjects with fused lumbar vertebrae, determined by X-rays and CT scans

SECONDARY OUTCOMES:
Device compliance | 6 months
  actual minutes per day device was used compared with prescribed treatment time
revision rate | 12 months
  how many subjects had to be reoperated (revised) at the same level(s) during the course of the study
SF-36 | 12 months
  used to assess the effect of PEMF treatment on subject quality of life
Oswestry Disability Index | 12 months
  used to examine the effect of PEMF treatment on subject disability
VAS pain | 12 months
  used to assess the effect of PEMF treatment on reduction of pain
EQ-5D | 12 months
  used to assess the effect of PEMF treatment on quality of life and economic impact

CONTACTS AND LOCATIONS:
Overall Officials: James T Ryaby, Ph.D., Principal Investigator — Orthofix Inc.
Locations (1):
- ClinTech Center for Spine Health, Johnstown, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
if we decide to share, we will only share deidentified summary data

REFERENCES:
- [Derived] Weinstein MA, Beaumont A, Campbell P, Hassanzadeh H, Patel V, Vokshoor A, Wind J, Radcliff K, Aleem I, Coric D. Pulsed Electromagnetic Field Stimulation in Lumbar Spine Fusion for Patients With Risk Factors for Pseudarthrosis. Int J Spine Surg. 2023 Dec 26;17(6):816-823. doi: 10.14444/8549. PMID 37884337